CLINICAL TRIAL: NCT04721730
Title: Prevention of Child Mental Health Problems in Southeastern Europe - Adapt, Optimize, Test, and Extend Parenting for Lifelong Health ' - 'RISE' - The Randomized Controlled Trial (Phase 3 of MOST)
Brief Title: Prevention of Child Mental Health Problems in Southeastern Europe - Phase 3
Acronym: RISE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Bremen (Other)
Collaborators: University of Klagenfurt (Other); University of Oxford (Other); Bangor University (Other); Babes-Bolyai University (Other); Institute for Marriage, Family and Systemic Practice - ALTERNATIVA (Other); Health for Youth Association, Moldova (Other); University of Cape Town (Other); Georgia State University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: H2020-779318-3; H2020-SC1-2017-RTD-779318 (Other Grant/Funding Number: European Commission)
Record Dates: First submitted 2021-01-13; First posted 2021-01-25 (Actual); Last update posted 2022-03-22 (Actual); Status verified 2022-03

CONDITIONS: Child Mental Disorder
Keywords: Parenting Programme
MeSH Terms: conditions — Neurodevelopmental Disorders

STUDY DESIGN:
Intervention Model Description: Participants will be randomly allocated 1:1 to the intervention group (5 sessions parent training "Parenting for Lifelong Health for Young Children"), and the control group (one lecture on parenting "Raising Healthy Children").
Who Masked: Outcomes Assessor
Masking Description: Participants will be allocated to groups after completion of pre-assessment. Thus, outcome assessors and participants will be blind to group allocation at pre-assessment. The implementation of the intervention will be conducted by different research staff (program coordinators and facilitators) than the assessments. Thus, data assessors are not aware of the group allocation of participants at the later assessment points (post, follow-up). To make sure that participants do not reveal their group allocation during the post- and follow-up assessment to the assessor, the data assessor will ask the participants to not share the group allocation at the beginning of the interview. Unblinding will only happen in case the participant reports a (serious) adverse event during the interview (at post- or follow-up assessment).
  Also, the data analysis team (Klagenfurt) will remain blind to group allocation, because the unrevealing of assignment will be done in Bremen.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- PLH-YC (Experimental): The Parents will receive the optimised version of the Parenting for Lifelong Health for Young Children from 2-9 y. (PLH-YC) identified in Phase 2.
  The groups will be conducted with 12 parents per group (with 2 facilitators). If local restrictions due to COVID-19 restrictions do not allow-in person meetings of this size, we will reduce the sample size (6 parents per group, and facilitator) and or conduct the groups online (e.g., using an online video software).
  For each session, parents will receive a snack (or food voucher of same amount), childcare, transportation support (if needed), and a certificate at the end. Also, parents participating in at least four out of five PLH sessions will get a small gift. If the groups need be conducted online because of the COVID-19 pandemic, the parents will receive pre-paid data or another voucher of the same amount.
  Interventions: Behavioral: PLH-YC
- Lecture (Active Comparator): Parents will receive a lecture called "Raising Healthy Children".
  The lecture will be conducted with 12 parents per group (with one facilitator). If local restrictions due to COVID-19 pandemic will not allow in-person meetings, the groups will be online (e.g., using a video meeting software).
  During the lecture, parents will receive a snack (or a food voucher of the same amount), childcare, transportation support (if needed), and a certificate at the end. If the lecture needs be conducted online because of the COVID-19 pandemic and associated restrictions, the parents will receive pre-paid data or another voucher of the same amount (instead of childcare, transport voucher and the snack).
  Interventions: Behavioral: Lecture

INTERVENTIONS:
Behavioral: PLH-YC — There will be 5 weekly 2-hour sessions. The optimised PLH-YC uses a participatory, non-didactic approach to engage parents. Parents learn positive parenting skills and how to manage child behaviour problems. The program includes Session 1: One-on-One Time and Say What You See, Session 2: Praise and Rewards, Session 3: Instructions, Redirect, Rules, and Routines, Session 4: Ignore and Consequences, Session 5: Reflection and Moving On. Core activities during sessions include group discussions illustrated vignettes, role-plays, collaborative problem solving, practicing skills at home.
  Other Names: Parenting for Lifelong Health for Young Children
  Arms: PLH-YC
Behavioral: Lecture — Lecture on parenting. This is a 26-slides power-point presentation that was developed by the University of Bremen for the purpose of this study. Duration: 1 to 1.5 hours. Content: 1) Stages of child development; (2) Potential risk factors for child emotional or behaviour problems; (3) Resources and protective factors; (4) Tips: What parents can do to promote children's development.
  Other Names: Raising Healthy Children
  Arms: Lecture

SUMMARY:
The overall RISE project aims to adapt, optimise and test a low-cost parenting programme for families in three southeastern European countries (North Macedonia, Republic of Moldova, Romania). Therefore, the investigators apply the Multiphase Optimization Strategy (MOST) and conduct the study over 3 phases: during the first Phase (Preparation) the feasibility of the intervention and the assessment and implementation procedures were tested in a small pilot study. In the second Phase (Optimization), 8 different programme combinations were tested in order to identify the most effective and cost-effective combination in the three countries. Now, in the third Phase (Evaluation), the optimised intervention identified in Phase 2 will be tested in a randomised controlled trial. The investigators also apply dimensions of the RE-AIM framework to maximise the reach, effectiveness, adoption, implementation within the existing service infrastructure and maintained use of the new intervention.

For the current Phase 3, the investigators aim to recruit a total of 864 parents (n = 288 per country) of children with elevated child behaviour problems aged 2 to 9 years. After pre-assessment the families will be randomly assigned to the intervention group or the control group. Parents in the intervention group will receive a parenting programme (5 sessions, Parenting for Lifelong Health for Young Children, PLH-YC) and the parents in the control condition will receive one lecture on parenting (Raising Healthy Children). Parents will be asked to complete assessments after intervention completion (post-assessment) and 12 months after pre-assessment (follow-up assessment) in order to detect immediate and more longterm effects.

DETAILED DESCRIPTION:
Over the past decade there have been increasing calls for the scale-up of evidence-based interventions in order to reduce the risk of violence against children in low- and middle-income countries (LMICs). In particular, group-based parenting programmes for families with young children have been shown to be effective in reducing the risk of child maltreatment and improving child wellbeing with promising evidence emerging from low- and middle-income countries. These group-based programmes typically aim to strengthen caregiver-child relationships through positive parenting and help parents to manage child behaviour problems through effective, age-appropriate, nonviolent discipline strategies.

Despite the emerging evidence of the effectiveness of parenting interventions in reducing violence against children, many local governments and service providers in LMICs face multiple challenges in implementing evidence-based parenting programmes in resource poor contexts. Parenting programmes are often too expensive to deliver effectively at scale in low-resource settings due to their complexity, intensity, and length. Parenting programmes developed and evaluated in other contexts also may not fit the local service delivery context and may require adaptation to be relevant to the local culture of families. Additional programme content may also be necessary to address acute economic deprivation, high community violence, and parental distress. The process of delivery may also need to be simplified to improve participant engagement and the quality of delivery.

As a result, it is essential that programmes implemented in LMICs are

* Effective at reducing violence against children,
* Integrated within the existing service delivery system of the country,
* Feasible and culturally acceptable to service providers and families, and
* Scalable in terms of their affordability, replicability, and sustainability while reaching a maximum number of beneficiaries.

However, there are currently very few parenting programmes that meet these criteria in LMICs (such as North Macedonia, Republic of Moldova, and Romania), where the need is the greatest.

The Parenting for Lifelong Health (PLH) initiative is focused on the development, evaluation, and dissemination of parenting programmes to reduce violence against children and improve child wellbeing in LMIC. It was established to address the need to develop low-cost, evidence-based parenting programmes that can be integrated within existing service delivery systems in LMIC. The PLH for Young Children from 2-9 y. (PLH-YC) programme includes general content like one-on-one time/child-led play; praising and rewarding children; instructions, household rules, and routines; managing difficult behaviours: ignore and consequences; reflection and moving on. Core activities during sessions include group discussions illustrated vignettes, role-plays, collaborative problem solving, practicing skills at home.

The overall RISE project has two general objectives: (1) the first objective relates to the adaption, optimisation and evaluation of selected best practice intervention condition (MOST), while (2) the second objective relates to implementation issues (RE-AIM).

The primary objective of the overall project is adapt, optimise and test a parenting programme so that it meets the specific needs and constraints of families in three LMIC in Southeastern Europe. The design is informed by the Multiphase Optimisation Strategy (MOST) and is conduced over 3 distinct phases: 1) Preparation, 2) Optimisation, and 3) Evaluation. In Phase 1, the feasibility of the intervention and research methods was tested in a small pilot study in North Macedonia, Republic of Moldova, and Romania. In Phase 2, 8 different programme components were tested in a factorial experiment to identify the most effective and cost-effective combination. In the present Phase 3, the optimised intervention (identified in Phase 2) will be tested in a randomised-controlled trial.

A secondary objective of this project is to carefully assess barriers to implementation, integration with existing service delivery systems, and scale-ups from the outset to facilitate sustainability and real world applicability at the end of the project. When introducing such an innovative intervention in resource-limited settings, it is important to focus on the implementation processes that increase reach, efficacy, adoption, and sustainability of culturally-adapted and optimized versions of the programme in addition to evaluating programme effectiveness. The theoretical model for the implementation framework in the RISE project is RE-AIM (Reach, Efficacy, Adoption, Implementation, Maintenance, Glasgow et al., 2011). As a result, investigators will examine the adoption (defined as the proportion of settings willing to initiate the intervention), reach (the proportion of eligible individuals that participate in the intervention) and implementation (the fidelity, adherence, dosage assessed with multiple measures) as well as on effectiveness and sustainability of the RISE project at the organizational and participants' level. In addition, it will be examined how implementation factors influence programme effectiveness, and how potential population characteristics might affect outcomes (e.g., moderators such as baseline parent mental health, for details see study protocol, Taut et al., in preparation).

The first two Phases have been successfully completed. For details of Phase 1, see trial registration (https://clinicaltrials.gov/ct2/show/NCT03552250) and study protocol (doi: 10.1136/bmjopen-2018-026684). For details of Phase 2, please refer to the trial registration (https://clinicaltrials.gov/ct2/show/NCT03865485) or the study protocol (https://doi.org/10.1016/j.cct.2019.105855).

This presently registered study relates to the Evaluation Phase (Phase 3). This randomised-controlled trial ist to test the effectiveness and the cost-effectiveness of the optimised intervention (identified in the factorial experiment, Phase 2) in the three LMIC North Macedonia, Republic of Moldova and Romania. More details can be found in the study protocol for Phase 3.

Note: The investigators have developed a stepwise safety plan in case the local restrictions due to COVID-19 pandemic will not allow in-person assessments and parent groups (as planned). The safety plan includes the reduction of the number of parents per group size switch to online delivery of PLH-YC and lecture / phone assessments. For more details, please see the study protocol (Taut et al., submitted).

Note: The investigators will assess further variables that are not mentioned in the outcome section. These are moderator variables that will be only assessed once (at baseline) and that are described in the study protocol (Taut et al., in preparation).

Note: Based on the experiences during the pre-assessments, an interim reduction of measures was necessary to prevent overburdening of families (more time needed for assessments because of the pandemic situation). It was decided to take out some of the other pre-specified outcome measures for the post-assessment (for details, see outcome section).

Note: Assessment of parent-child relationship: In addition to the coherence rating, two scales of the FAARS rating (Warmth, Criticism) were added for the following reasons: The FAARS scales are assumed to be closely related to the mechanisms and outcomes of a social learning theory based parenting program and may better capture the expected change. These scales also showed good validity in other parenting intervention studies (e.g., Smith et al., 2013).

ELIGIBILITY:
Inclusion Criteria (for caregivers/parents):

1. Age 18 or older;
2. Primary caregiver responsible for the care of a child between the ages of two and nine;
3. Report elevated levels of child behavior problems for the child that he/she chooses to be part of the study (based on the Child and Adolescent Disruptive Behavior Inventory, oppositional defiant disorder subscale (8 items); scores of 10 or more
4. Have lived in the same household as this child at least four nights a week in the previous month and will continue to do so;
5. Agreement of being randomized to one of the two conditions
6. Provision of Informed consent to participate in the full study
7. Language skills to participate in the group/lecture (e.g., with someone that helps with the translation).

Exclusion Criteria (for caregivers/parents):

1. Parents with legal restriction to child care - indirectly assessed via the inclusion criterion on the number of nights/day with the child/per week

Inclusion Criteria (for facilitators of PLH/lecture):

1. Age 18 or older;
2. Participate in PLH facilitator training workshop /lecture training workshop;
3. Agreement to either deliver the lecture (one session) or PLH-YC (five sessions);
4. Provision of consent to participate in the full study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 823 (Actual)
Dates: Start 2020-12-07 (Actual); Primary Completion 2022-03-14 (Actual); Study Completion 2022-03-14 (Actual)

PRIMARY OUTCOMES:
Change in level of aggressive behaviour in children: Child Behavior Checklist (CBCL) 11/2-5 and 6-18, parent-report, sub-scale "Aggressive behaviour" (with 19 items (CBCL ½ - 5) and 18 items (CBCL 6-18), continuous sub-scale score | pre: Jan/Feb 2021; post: approx. 4 months after pre assessment (May/June 2021); follow-up: approx. 10 -12 months after pre-assessment (Dec 2021 - Feb 2022)
  The primary outcome child oppositional aggressive behaviour is assessed with 3 indicators: 1) parent-report: The CBCL is part of the Achenbach System of Empirically Based Assessment (ASEBA) and is available for different age ranges, including the targeted range in the present study. For Phase 3, the parent-report versions for children aged 1½-5 and 6-18 are employed. The aggressive behaviour sub scale (CBCL ½ - 5 version: 19 items, CBCL 6-18: 18 items) belongs to the externalising scale and assesses aggressive behaviour (e.g., "Argues a lot"). The total raw score ranges from 0 to 38 in the CBCL ½ - 5 version and 0-36 in the CBCL 6-18 version, with higher scores indicating more aggressive child behaviour. Items are rated on a 3-point Likert scale (2 = very true or often true of the child; 0 = not true of the child).
Change in prevalence of Externalising Disorders in Children (MINI-KID), binary total score | pre: Jan/Feb 2021; post: approx. 4 months after pre assessment (May/June 2021); follow-up: approx. 10 -12 months after pre-assessment (Dec 2021 - Feb 2022)
  The primary outcome child oppositional aggressive behaviour is assessed with 3 indicators: 2) clinical interview: The Mini International Neuropsychiatric Interview for Children and Adolescents - Parent Version (MINI-KID-P) will be used to assess whether the criteria for a) Conduct Disorder (CD) or b) Oppositional Defiant Disorder (ODD) are met (yes/no). The results of the two disorders will be combined to one binary total score with 0 = no externalising disorder and 1 = current externalising disorder (ODD or CD).
Change in Parent Daily Ratings (PDR): oppositional and aggressive sub scale (12 items), continuous sub-scale score | PLH group: after the first, third and fifth session. lecture: after the lecture, 2 and 4 weeks later
  The primary outcome child oppositional aggressive behaviour is assessed with 3 indicators: 3) daily reports: The PDR oppositional and aggressive sub-scale (10 items) and 2 positive items will be used to monitor child behavioral problems. We excluded the last item from the scale ("he/she pouts") because this question caused translation problems in the three implementation countries during the last assessment. The item was not understood correctly by parents and assessors and thus did not result in valid answers. Parent will report on their child's behaviour within the last 24 hours (answer format: did occur/did not occur). The oppositional and aggressive subscale mean score will be calculating (score range: 0-1) with higher scores indicating more child problem behaviour within the last 24 hours. Additional exploratory analyses will include the mean score of the two positive items (range: 0 -1) with higher values indicating more frequent positive child behaviour.

SECONDARY OUTCOMES:
Change in level of internalising problem behaviour in children: Child Behavior Checklist (CBCL) 11/2-5 (31 items) and 6-18 (32 items) parent-report, Internalizing Scale; continuous sub-scale score | pre: Jan/Feb 2021; post: approx. 4 months after pre assessment (May/June 2021); follow-up: approx. 10 -12 months after pre-assessment (Dec 2021 - Feb 2022)
  The CBCL is part of the Achenbach System of Empirically Based Assessment (ASEBA) and is available for different age ranges, including the targeted range in the present study. For the present study, the parent-report versions for children aged 1½ - 5 and 6-18 are employed. It is the most widely used instrument for assessing child behavioral and emotional symptoms. In addition to the possibility to separate behavioral from emotional symptoms, the CBCL allows for assessment in multiple languages, including Romanian (all ages), Russian (all ages), and Macedonian (6-18 version). It is a very well validated instrument that has been used across different prevention and treatment studies. The internalising subscale raw score ranges from 0 to 62 (CBCL/1 ½ - 5 version) and 0 to 64 (CBCL/ 6 - 18 version) with higher scores indicating more emotional problems.
Change in frequency of dysfunctional parenting: Parenting Scale (PS) / self-report (shortened version); continuous total score and 2 sub-scale scores | pre: Jan/Feb 2021; post: approx. 4 months after pre assessment (May/June 2021); follow-up: approx. 10 -12 months after pre-assessment (Dec 2021 - Feb 2022)
  This measure is widely used in parenting interventions across the world. The scale was designed to explicitly measure dysfunctional discipline practices in parents. Three subscales may be derived (Laxness, Overreactivity, and Verbosity). For phase 3, the subscale Verbosity is excluded due to poor performance in the pilot study, consistent with numerous other studies evaluating this subscale's psychometric properties. Each item is rated on a 7-point Likert Scale in which parents are presented with a situation and then are asked to choose between two alternative responses to a situation (1 = most effective; 7 = most ineffective; i.e., situation: "When I say my child can't do something"). For computation of the subscale scores as well as the total score, the responses on the items are averaged. We will use a modified total score (only from two subscales Laxness & Overreactivity).
Change in frequency of positive parenting and effective discipline: Parenting of Young Children Scale (PARYC) / self-report (21 items); continuous total score | pre: Jan/Feb 2021; post: approx. 4 months after pre assessment (May/June 2021); follow-up: approx. 10 -12 months after pre-assessment (Dec 2021 - Feb 2022)
  Positive parenting behavior will be assessed using parent-report of the Parenting of Young Children Scale (PARYC, 21 items). The PARYC measures the frequency of parent behaviour over the previous month. Items are summed to create a total frequency scores parenting behaviour as well as for the sub-scales: positive parenting (7 items, e.g., "how often do you play with your child"), setting limits (7 items, e.g., "how often do you stick to your rules and not change your mind") and proactive parenting (7 items, e.g., "how often do you explain what you want your child to do in clear and simple ways"). This scale has been used in PLH trials in other countries and will allow comparison of results to those studies.
Change in daily report of effective parenting behaviour (5 items of Alabama Parenting Questionnaire), continuous score | PLH group: after the first, third and fifth session. lecture: after the lecture, 2 and 4 weeks later
  We will use 5 items from the Alabama Parenting Questionnaire phone interview (3 items for positive and 2 for negative parent behaviours) to assess daily reports of parenting behavior. The original answer format was adapted to fit the PDR format (0=did occur/1=did not occur). One overall mean score will be calculated (ranging from 0 to 1) with higher scores indicating more effective parenting behaviour (ineffective parenting items will be reverse-scored).
Change in parent-child relationship quality as measured via FMSS (Five Minute Speech Sample) coherence; continuous total score | pre: Jan/Feb 2021; post: approx. 4 months after pre assessment (May/June 2021); follow-up: approx. 10 -12 months after pre-assessment (Dec 2021 - Feb 2022)
  The FMSS assesses the caregiver's attitudes and feelings about the child and his/her perceptions of the quality of their relationship. The parent is instructed to talk about his/her child for five minutes. The parent-report is audio-recorded and rated by trained coders. The overall coherence scale ranges from 1 (not coherent picture of child) to 7 (very coherent picture of child) with higher scores indicating a more coherent narrative which indicates a better parent-child relationship. If inter-rater reliability of sub-scales is fair enough (ICC of .70 or higher), additional exploratory analyses will comprise the sub-scales concern / worry (1 "no worry and concern" to 7 "thematic concern and worry"), acceptance and warmth vs. rejection (1 "strong rejection" to 7 "high warmth and acceptance"), and separateness (1 "no clear separation" to 7 "complete separateness"; incl. boundary dissolution (BD) answer format: 0, 1, 2 with higher scores indicating more BD).
Change in parent-child relationship quality as measured via FMSS (Five Minute Speech Sample) Family Affective Attitude Rating Scale (FAARS), sub scales Warmth and Criticism; continuous total score | pre: Jan/Feb 2021; post: approx. 4 months after pre assessment (May/June 2021); follow-up: approx. 10 -12 months after pre-assessment (Dec 2021 - Feb 2022)
  The FMSS assesses the caregiver's attitudes and feelings about the child and his/her perceptions of the quality of their relationship. The parent is instructed to talk about his/her child for five minutes. The parent-report is audio-recorded and rated by trained coders. Parents are rated using two sub scales of the FAARS on 9-point Likert items ranging from 1 "no evidence for the duration of the speech sample" to 9 "two or more concrete, unambiguous examples of a particular behaviour or attribute" on each of 5 items per sub scale. Sub scale scores (mean of items): For the Criticism sub scale, higher scores indicate more negative attitudes (and thus a lower parent-child relationship quality); while higher scores on the Warmth sub scale indicate more positive attitudes (and thus a better relationship quality).
Change in frequency and incidence of child maltreatment: ISPCAN-Child Abuse Screening Tool-Intervention (ICAST-I)/ self-report (16 items); main focus on continuous total score, 2nd question: any effect of intervention on any of the 3 sub-scale score | pre: Jan/Feb 2021; post: approx. 4 months after pre assessment (May/June 2021); follow-up: approx. 10 -12 months after pre-assessment (Dec 2021 - Feb 2022)
  Child maltreatment (CM) will be measured using parent report of the ICAST-I, an adaptation of an instrument measuring parent-report of child abuse and neglect (ICAST-TC, Trial Children). The ICAST-TC measures four types of abuse: physical, emotional and sexual abuse, as well as neglect. The response code was adapted to a scale from 0 to more than 8 times to assess the frequency of a certain behaviour in the past month. This study will assess incidence of CM by creating dichotomous variables for physical abuse, verbal abuse, and neglect, as well as an overall indication of previous child abuse. We will also assess frequency of overall abuse by summing all of the subscales as well as for each individual subscale. Regarding emotional abuse, a 5-item-version is used. Sexual abuse is not assessed.
  If assessments cannot take place in-person (due to COVID-19 restrictions), this measure will not be administered during the phone assessment because of the sensitive nature of items.
Change in levels of psychological distress in parents: Depression, Anxiety, and Stress Scales - short version/ self-report (21 items); continuous total score | pre: Jan/Feb 2021; post: approx. 4 months after pre assessment (May/June 2021); follow-up: approx. 10 -12 months after pre-assessment (Dec 2021 - Feb 2022)
  Depression, Anxiety, Stress Scales (DASS) will assess parent-report of psychological distress in parents, a 21-item scale used as a screening tool to measure depression, anxiety, and stress in adults. Caregivers report on the frequency of symptoms in the previous week using a Likert scale (0 = Never, 1 = Sometimes, 2 = Often, 3 = Always; e.g., "I felt that I had nothing to look forward to"). Total DASS scores range from 0 to 63 with subscales from 0 to 21. The DASS is a widely used measure across parenting studies including those of PLH-YC and will allow comparison to existing results of intervention studies in non-LMICs.
Change in levels of parenting stress: Parenting Stress Scale (18-items); continuous total score | pre: Jan/Feb 2021; post: approx. 4 months after pre assessment (May/June 2021); follow-up: approx. 10 -12 months after pre-assessment (Dec 2021 - Feb 2022)
  The Parental Stress Scale measures parental stress across different domains (rewards, stressors, satisfaction, loss of control) with 18 items. An example, from the domain stressors, is "The major source of stress in my life is my child(ren)". Caregivers answer on a scale from strongly disagree (1) to strongly agree (5). The overall score ranged from 18 to 90 with higher scores indicating more parental stress.
Change in levels of parental relationship quality: Couple Satisfaction Index / self-report (4 items); continuous total score | pre: Jan/Feb 2021; post: approx. 4 months after pre assessment (May/June 2021); follow-up: approx. 10 -12 months after pre-assessment (Dec 2021 - Feb 2022)
  This 4-item measure assesses relationship satisfaction among intimate partners. Items are summed to create a total score. CSI-4 scores can range from 0 to 21. Higher scores indicate higher levels of relationship satisfaction. CSI-4 scores falling below 13.5 suggest notable relationship dissatisfaction.
Change in levels of Intimate Partner Violence (29 items); continuous total score and 4 sub-scales (level of severity) | pre: Jan/Feb 2021; post: approx. 4 months after pre assessment (May/June 2021); follow-up: approx. 10 -12 months after pre-assessment (Dec 2021 - Feb 2022)
  Intimate partner violence will be assessed with a screening instrument, the family maltreatment measure (Heyman et al. 2013) and an adaption of the revised Conflict Tactics Scale (CTS2S). The measure assesses adult self-report of perpetration and victimisation of intimate partner aggression. Assessments measure the frequency of negotiation, physical assault, psychological aggression, and physical injury. This measure indicates an overall indication of IPV on a level of severity (sum of items) and prevalence (dichotomous variable indicating experience of conflict or not) as well as for each subscale. Only severity is examined here. For the current study a 9-point Likert scale of 0 to 8 is used, with an additional response for incidences that happened but not in the past month.
  If assessments cannot take place in-person (due to COVID-19 restrictions), this measure will not be administered during the phone assessment.
Change in Child Quality of Life: Child Health Utility 9D (CHU9D; 9 items); continuous total score | pre: Jan/Feb 2021; post: approx. 4 months after pre assessment (May/June 2021); follow-up: approx. 10 -12 months after pre-assessment (Dec 2021 - Feb 2022)
  The CHU9D measures parent-reported child health-related quality of life. The questionnaire consists of nine dimensions (worried, sad, pain, tired, annoyed, schoolwork/homework, sleep, daily routine, activities) with five levels (e.g., 1 = "don't feel worried"; 5 = "very worried"). Higher scores indicate lower levels of quality of life. The scores of the CHU9D range from 9-45.
RE-AIM Reach: Enrollment rate | approx. 4 months after pre-assessment (May/June 2021)
  Total number of caregivers who attend the first session of the PLH/ the lecture group divided by the number of families recruited in that condition).
RE-AIM Reach: Participation rate | approx. 4 months after pre-assessment (May/June 2021)
  Only for caregivers that were allocated to the PLH condition: percentage of sessions attended out of the 5 sessions

OTHER OUTCOMES:
RE-AIM Implementation: Fidelity Lecture | approx. 4 months after pre-assessment (May/June 2021)
  Percentage of session activities delivered per session: The number of total activities actually implemented (yes/no), divided by the number of session activities (assessed via a facilitator checklist, n = 22 activities).
RE-AIM Implementation: Fidelity PLH programme | approx. 4 months after pre-assessment (May/June 2021)
  Percentage of session activities delivered per session: The number of total activities actually implemented (yes/no), divided by the number of session activities by facilitator(assessed via a facilitator checklist, n = 22 activities).
RE-AIM Implementation: Quality of delivery PLH | approx. 4 months after pre-assessment (May/June 2021)
  PLH-Facilitator Assessment Tool (PLH-FAT): Seven standard behavior categories are grouped into two scales based on the core activities and process skills. Assessment of core activities includes quality of delivery during home activity review, illustrated story discussions, and practicing skills. Assessment of process skills includes modeling skills, collaborative facilitation approach, encouragement of participation, and leadership skills.
RE-AIM Implementation: Quality of delivery lecture | approx. 4 months after pre-assessment (May/June 2021)
  The delivery skills of the facilitators will be assessed with one overall quality of delivery item (0 = inadequate, 4 = excellent) which will be rated by trained coders.
Cost-effectiveness / cost-analyses - CBCL (Child Behavior Checklist (CBCL) 11/2-5 and 6-18, parent-report) sub-scale "Aggressive behaviour" (with 19 items (CBCL ½ - 5) and 18 items (CBCL 6-18) | approx. 4 months after pre assessment (May/June 2021); follow-up: approx. 10 -12 months after pre-assessment (Dec 2021 - Feb 2022)
  Cost-effectiveness ratio in terms of Euros per 1 point reduction of the CBCL aggressive sub-scale score of the PLH 2-9 program.
  The CBCL aggressive sub-scale score ranges from 0 to 38 in the CBCL ½ - 5 version and 0-36 in the CBCL 6-18 version, with higher scores indicating more aggressive child behaviour.
Cost-effectiveness / cost-analyses - Parenting Scale (PS) | approx. 4 months after pre assessment (May/June 2021); follow-up: approx. 10 -12 months after pre-assessment (Dec 2021 - Feb 2022)
  Cost-effectiveness ratio in terms of Euros per 1 point reduction of the Parenting Scale (total score) score of the PLH 2-9 program.
  For the parenting scale, a modified total score (only from two sub-scales Laxness & Overreactivity) will be used. For computation of this modified total score, the responses on the items are averaged, ranging from 1 to 7. Higher scores indicate more dysfunctional parenting behaviour.
Cost-effectiveness / cost-analyses - Parenting of Young Children Scale (PARYC) | approx. 4 months after pre assessment (May/June 2021); follow-up: approx. 10 -12 months after pre-assessment (Dec 2021 - Feb 2022)
  Cost-effectiveness ratio in terms of Euros per 1 point reduction of the Parenting of Young Children Scale (PARYC, 21 items) (total score) score of the PLH 2-9 program.
  For the PARYC total frequency score, the 21 items are summed ranging from 21 to 147 with higher scores indicating more positive parenting behaviour and effective discipline.
Cost-effectiveness / cost-analyses - Child Quality of life (Child Health Utility 9D, CHU9D; 9 items) | approx. 4 months after pre assessment (May/June 2021); follow-up: approx. 10 -12 months after pre-assessment (Dec 2021 - Feb 2022)
  Cost-effectiveness ratio in terms of Euros per 1 point reduction of the child quality of life (Child Health Utility 9D) (total score) score of the PLH 2-9 program.
  The total score of the CHU9D ranges from 9-45. Higher scores indicate lower levels of quality of life.
Child and Adolescent Behavior Inventory (CABI), oppositional defiant disorder sub scale (9 items); continuous sub-scale score | pre: Jan/Feb 2021
  The CABI questionnaires assesses different types of problem behaviour in childhood and adolescence. The CABI exists of 75 items measuring different areas of psychopathology, e.g., anxiety, depression, conduct disorder or attention deficit hyperactive disorder. Eight items assess oppositional defiant disorder directed towards adults and one additional item measures if any of the eight behaviors currently cause significant problems. The sum score of the first eight items can range from 0-40 and will be used as eligibility screening tool. Respondents with scores ≥10 will be included in the study. Higher scores indicate higher levels of symptoms. In addition, the sum score will be used as an outcome measure for the secondary caregivers (assessed at pre, post, follow-up).
Change in prevalence of ADHD (Mini International Neuropsychiatric Interview for Children and Adolescents - Parent Version); binary total score | pre: Jan/Feb 2021; post: approx. 4 months after pre assessment (May/June 2021); follow-up: approx. 10 -12 months after pre-assessment (Dec 2021 - Feb 2022)
  The MINI-KID-P (structured clinical interview, parent report version) will be employed to assess whether or not the criteria for ADHD (F90.0, F90.1) are currently met (yes/no). The results will be combined to one binary total score 0 (no ADHD) and 1 (current ADHD, criteria met).
Change in Couple Conflict (10 items); continuous total score. | pre: Jan/Feb 2021; post: approx. 4 months after pre assessment (May/June 2021); follow-up: approx. 10 -12 months after pre-assessment (Dec 2021 - Feb 2022)
  For respondents who are in a romantic relationship, overt conflict between couples as observed by the child will be assessed using the O'Leary Porter Scale (OPS; Porter & O'Leary, 1980). This measure assesses adult self-report of hostile couple conflict as witnessed by the child. Assessments measure the frequency of hostility, including quarrels, sarcasm, and domestic violence in front of the child (sum of items). Answers are coded on a 5-point Likert scale of 1 (Never) to 5 (Very often). Thus, the score ranges from 10 to 25 with higher scores indicating more overt couple conflict.
Change in Coparenting Quality (10 items); continuous total score and 2 subscales. | pre: Jan/Feb 2021; post: approx. 4 months after pre assessment (May/June 2021); follow-up: approx. 10 -12 months after pre-assessment (Dec 2021 - Feb 2022)
  For respondents who coparent their child with another caregiver, coparenting quality will be assessed using two subscales of the Coparenting Relationships Scale (CRS; Feinberg et al., 2012), Coparenting Agreement (4 items) and Coparenting Undermining (6 items). This measure assesses adult self-report of coparenting quality between them and their coparent. Answers are coded on a 7-point Likert Scale from 0 (Not true of us) to 6 (Very true of us). The mean of the Coparenting Agreement subscale ranges from 0-6 with higher scores indicated greater coparenting agreement. The mean of the Coparenting Undermining subscale ranges from 0-6 with higher scores indicating more coparenting undermining. These scales are also combined, after reversing the undermining items, for an overall coparenting quality mean ranging from 0-6, with higher scores indicating better coparenting quality.
Change in Parental Self-Regulation (1 item), continuous core | pre: Jan/Feb 2021; post: approx. 4 months after pre assessment (May/June 2021); follow-up: approx. 10 -12 months after pre-assessment (Dec 2021 - Feb 2022)
  Parental Self-Regulation will be assessed using The Pause item. This measure assesses adult self-reported ability to pause before reacting reflexively to negative child behaviors. This assessment measures the frequency of parents taking a moment to think or calm down before reacting when he or she feels upset or stressed with the child. Answers are coded on a 4-point Likert scale of 0 (Never) to 3 (Very often) with higher scores reflecting better self-regulation ability of parents.
Change in Frequency and Quality of Family Dinner (4 items); continuous total score and 2 sub-scales. | pre: Jan/Feb 2021; follow-up: approx. 10 -12 months after pre-assessment (Dec 2021 - Feb 2022)
  Family dinner will be assessed using the Family Dinner Scale (FDS; Fishel, 2020). This measure assesses adult self-reported frequency and quality of family dinners. Assessments first measure the frequency of family dinner, and if the family has dinner together at least rarely, the quality of their dinners is then assessed (conversation, positive affect, reducing distractions). Answers are coded on a 4-point Likert scale of 1 (Never) to 4 (Often). This measure indicates the overall quality of family dinners (mean of all items ranging from 0 to 4 with higher scores indicating better quality family dinners), and frequency (item 1 ranging from 0-4) and quality (items 2-4, means ranging from 0-4) can also be examined separately.
Change in levels of social community support, MOS Social Support Survey - Emotional Support Sub-scale (8 items); continuous sub-scale score | pre: Jan/Feb 2021; follow-up: approx. 10 -12 months after pre-assessment (Dec 2021 - Feb 2022)
  Perceived social support will be measured using the emotional support subscale of the Medical Outcome Study Social Support Survey (MOS-SSS, 8-items). In validation studies this scale has shown excellent internal consistency (α = 0.91 to 0.97) and test-retest reliability (α = 0.72 to 0.78). Parents report on the frequency of how often they receive emotional support (e.g., "someone you can count on to listen to when you need to talk") on a Likert-like scale of 1 to 5 (1 = none of the time; 5 = all of the time). Total scores are calculated by averaging the scores for each item and then transformed into a 0 to 100 scale. The scale was found to be distinct from related health measures, which is important for the present study.
Change in alcohol misuse: Alcohol Use Disorders Identification Test AUDIT-C, 3 items), continuous total score | pre: Jan/Feb 2021; follow-up: approx. 10 -12 months after pre-assessment (Dec 2021 - Feb 2022)
  The Alcohol Use Disorders Identification Test - Consumption (AUDIT-C) is a modified version of the 10-item AUDIT instrument that was developed by the WHO. It is a 3-item alcohol screener that reliably identifies patients who are hazardous drinkers or have active alcohol use disorders (Bush, Kivlahan & McDonell, 1989). Each item asked about the frequency of a particular behavior, using a 5-point Likert Scale. Items were then summed up to build a total AUDIT-C score on a scale from 0 to 12." Response options range from 0 (Never;1 or 2) to 4 (4 or more times a week, 10 or more; Daily or almost Daily). Higher scores indicate more alcohol use.
Change in Participant's General Health (6 items incl. 3 items from the Medical Outcomes Study (MOS) Short Form-12 Health Survey (SF-12)), 3 continuous sub-scale scores | pre: Jan/Feb 2021; follow-up: approx. 10 -12 months after pre-assessment (Dec 2021 - Feb 2022)
  Caregiver general health will be assessed using three items from the Medical Outcomes Study (MOS) Short Form-12 Health Survey (SF-12). This scale is an adapted version of the MOS SF-34 Health Survey. Items include difficulty in normal daily activities, such as cleaning the home, going to work, or carrying a child. Response options are based on a 3-point Likert-like scale (1 = yes, limited a lot; 3 = no, not limited at all). The third item requires respondents to assess their overall health on a 5-point Likert scale (1 = excellent; 5 = poor). Three additional items ask respondents whether they or their child have a (physical or mental) disability. If they respond yes, they are asked to specify which type of disability. Calculated scores include parental health (sum of items 1 to 3), parental health including disabilities (sum of items item 1-4), and child health including disabilities (sum of items 5 and 6).

CONTACTS AND LOCATIONS:
Overall Officials: Nina Heinrichs, Prof., Principal Investigator — University of Bremen; Heather Foran, Prof., Principal Investigator — University of Klagenfurt; Jamie Lachman, Dr., Principal Investigator — University of Oxford; Adriana Baban, Prof., Principal Investigator — Babes-Bolyai University; Marija Raleva, Prof., Principal Investigator — Institute for Marriage, Family and Systemic Practice - ALTERNATIVA; Galina Lesco, Dr., Principal Investigator — Health for Youth Association, Moldova; Frances Gardner, Prof., Principal Investigator — University of Oxford; Judy Hutchings, Prof., Principal Investigator — Bangor University; Catherine Ward, Prof., Principal Investigator — University of Cape Town; Xiangming Fang, Prof., Principal Investigator — Georgia State University
Locations (3):
- Health for Youth Association, Chisinau, MD, Moldova
- Institute for Marriage, Family and Systemic Practice - ALTERNATIVA, Skopje, North Macedonia
- Babes Boylai University, Cluj-Napoca, Romania

IPD SHARING:
Plan to Share IPD: Yes
It is planned to share results to members of the scientific community with an interest in parenting interventions, behavioral problems in children, process evaluation, the transferability of interventions across cultures and contexts, and the MOST (the Multiphase Optimization Strategy). The aim is to sustain the intervention after the end of the project by including local authorities, policy makers, and other stakeholders such as community groups and caregivers in the intervention from each country. Further, we will archive the dataset and upload metadata in the certified repository Zenodo at https://zenodo.org/. Further details about IPD Sharing are described in the Data Management Plan and this is available by contacting Prof. Heather Foran (heather.foran@aau.at).
Supporting Information: Study Protocol, SAP, ICF
Time Frame: at the end of the project

REFERENCES:
- [Background] Frantz I, Foran HM, Lachman JM, Jansen E, Hutchings J, Baban A, Fang X, Gardner F, Lesco G, Raleva M, Ward CL, Williams ME, Heinrichs N. Prevention of child mental health problems in Southeastern Europe: a multicentre sequential study to adapt, optimise and test the parenting programme 'Parenting for Lifelong Health for Young Children', protocol for stage 1, the feasibility study. BMJ Open. 2019 Jan 25;9(1):e026684. doi: 10.1136/bmjopen-2018-026684. PMID 30782760
- [Background] Lachman JM, Heinrichs N, Jansen E, Bruhl A, Taut D, Fang X, Gardner F, Hutchings J, Ward CL, Williams ME, Raleva M, Baban A, Lesco G, Foran HM. Preventing child mental health problems through parenting interventions in Southeastern Europe (RISE): Protocol for a multi-country cluster randomized factorial study. Contemp Clin Trials. 2019 Nov;86:105855. doi: 10.1016/j.cct.2019.105855. Epub 2019 Oct 24. PMID 31669446
- [Background] Taut D, Baban A, Frantz I, Danila I, Lachman JM, Heinrichs N, Ward CL, Gardner F, Fang X, Hutchings J, Raleva M, Lesco G, Murphy H, Foran H. Prevention of child mental health problems through parenting interventions in Southeastern Europe (RISE): study protocol for a multi-site randomised controlled trial. Trials. 2021 Dec 27;22(1):960. doi: 10.1186/s13063-021-05817-1. PMID 34961518
- [Derived] Frantz I, Foran HM, Lachman JM, Gardner F, McMahon RJ, Ogden T, Hutchings J, Costin MR, Kunovski I, Raleva M, Mueller J, Heinrichs N. Adverse event assessment in a parenting programme: experiences from a multisite randomised controlled trial. Trials. 2024 Aug 17;25(1):547. doi: 10.1186/s13063-024-08357-6. PMID 39154169
- See also: Trial Registration Phase 1 — https://clinicaltrials.gov/ct2/show/NCT03552250
- See also: Trial Registration Phase 2 — https://clinicaltrials.gov/ct2/show/NCT03865485